CLINICAL TRIAL: NCT00741832
Title: The Effects of a Positive Expiratory Pressure (PEP) on Dyspnea and Dynamic Hyperinflation During Exercise in COPD Patients
Brief Title: The Effects of a Positive Expiratory Pressure (PEP) on Dyspnea and Dynamic Hyperinflation During Exercise in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Graduate School, Khon Kaen university
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: KKU-4950900021
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; dynamic hyperinflation; dyspnea; recovery; positive expiratory pressure; exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): Patients breath while a conical positive expiratory pressure device during exercises
  Interventions: Device: Conical Positive Expiratory Pressure Device (C-PEP)
- C (Active Comparator): Patients (normal) breath during exercise
  Interventions: Other: Control breathing

INTERVENTIONS:
Device: Conical Positive Expiratory Pressure Device (C-PEP) — Conical positive expiratory pressure device (C-PEP) in this study was designed on the principle of expiratory flow retardation. The principle occurs when exhaling through a small tube diameter, i.e. a small straw, pursed lip breathing, or positive expiratory pressure. Expiratory retardation, results from a decrease in tube diameter, creates flow resistance during exhalation. With flow resistance, the greater the flow the greater the back pressure, and the less the flow the lower the pressure. Expiratory retardation was applied in an attempt to facilitate exhalation and to relieve the air trapping.
  The optimal design was found to be: cone shape, proximal diameter is 2.0 cm, distal diameter is 0.6 cm, and length is 2.5 cm.
  Subjects will rest for 10-15 minutes until HR, BP are stabilized. They will undertake 15 min of alternating quadriceps exercise (30% 1 RM) either breathing with the C-PEP device.
  Arms: I
Other: Control breathing — Subjects will rest for 10-15 minutes until HR, BP are stabilized. They will undertake 15 min of alternating quadriceps exercise (30% 1 RM) either breathing normally.
  Arms: C

SUMMARY:
From the relationship between pathophysiology of chronic obstructive pulmonary disease (COPD), dyspnea, and dynamic hyperinflation during ventilatory increasing, the investigators hypothesize that

1. Positive expiratory pressure (PEP) breathing will reduce dyspnea more than normal breathing during exercise in mild to moderate COPD patients.
2. PEP breathing will improve dynamic hyperinflation during exercise more than normal breathing in mild to moderate COPD patients.
3. PEP breathing will improve cardiorespiratory function during exercise than normal breathing in mild to moderate COPD patients.

DETAILED DESCRIPTION:
Expiratory airflow limitation is the pathophysiological hallmark of chronic obstructive pulmonary disease (COPD) that leads to air trapping and increases in dynamic hyperinflation (DH) and consequently causes dyspnea during exercise. Although pursed lips breathing is a simple technique that provides a positive back pressure may retard the airway collapsed, but previous studies showed an unsuccessful reduction of DH which might cause by insufficient back pressure. And thereby a conical positive expiratory pressure (C-PEP) has been developed in our laboratory to generate back pressure higher than pursed lips breathing. Moreover, an effect of PEP on DH has not carried out in patient with COPD. Therefore, the objective of the present study was to examine effects of a C-PEP on DH and respiratory response during exercise in patient with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable mild-to-moderate COPD (Both stages: FEV1/FVC < 70%. Mild stage: FEV1 ≥ 80% predicted; Moderate stage: 50% ≤ FEV1 < 80% predicted according to Global Initiative Obstructive Lung Disease (GOLD) guideline).
* Free of exacerbations for more than 4 weeks (as defined by a change to pharmacological therapy, admission to hospital or ER or unscheduled clinic visit).
* Good communication

Exclusion Criteria:

* Older than 70 years old
* Musculoskeletal problems that limit mobility
* Cardiovascular disease
* Neurological or psychiatric illness
* Patient on long term oxygen or domiciliary noninvasive positive pressure ventilation
* Any other comorbidities which would affect ability to undertake exercise test

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Inspiratory Capacity | at 0th, 5th, ~20th minutes of exercises
Borg scale | at 0th and 20th minutes of exercises

SECONDARY OUTCOMES:
Heart Rate | every minutes of exercise and recovery periods
Exercise time | at the times when participants stop exercises
Recovery time | the periods between end of symptomatic limited constance workload exercises to full recovery heart rate
Respiratory rate | every minutes of exercise and recovery periods
Inspiratory time | every minutes of exercise and recovery periods
Expiratory time | every minutes of exercise and recovery periods
Sp02 | every minutes of exercise and recovery periods
PetCO2 | every minutes of exercise and recovery periods
Mouth pressure | every minutes of exercise periods
Flow rate | every minutes of exercise periods

CONTACTS AND LOCATIONS:
Overall Officials: Watchara Boonsawat, Philosophy, Study Director — Department of medicine, Faculty of medicine, Khon Kaen university; Tadsawiya Padkao, Bachelor, Study Chair — Physical Therapy department, Faculty of Associated Medical Sciences, Khon Kaen university; Chulee CU Jones, Philosophy, Study Director — Phusical Therapy Department, Faculty of Associated Medical Sciences, Khon Kaen university, Thailand
Locations (1):
- Pulmonary research room of physical therapy department, Faculty of associated medical sciences, Khon Kaen university, Khon Kaen, Changwat Khon Kaen, Thailand

REFERENCES:
- [Derived] Padkao T, Boonsawat W, Jones CU. Conical-PEP is safe, reduces lung hyperinflation and contributes to improved exercise endurance in patients with COPD: a randomised cross-over trial. J Physiother. 2010;56(1):33-9. doi: 10.1016/s1836-9553(10)70052-7. PMID 20500135